CLINICAL TRIAL: NCT01554098
Title: A Comparison of Two Colonoscopic Withdrawal Techniques on Colonic Polyp Detection: an Open, Randomised, Cross Over Trial
Brief Title: A Comparison of Two Colonoscopic Withdrawal Techniques
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: STH16220
Record Dates: First submitted 2012-02-27; First posted 2012-03-14 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Intestinal Polyps
Keywords: Polyp detection; Supine; Colonoscope withdrawal; Patient position; Dynamic position change
MeSH Terms: conditions — Intestinal Polyps; Deception | interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strategy : supine first (Active Comparator): This study will be performed as a cross over study, comparing withdrawal in the supine position versus withdrawal with dynamic position change.
  Withdrawal in supine position followed by withdrawal with dynamic position change
  Interventions: Procedure: Strategy : Supine first
- Strategy : dynamic first (Active Comparator): This study will be performed as a cross over study, comparing withdrawal in the supine position versus withdrawal with dynamic position change.
  Interventions: Procedure: Strategy : dynamic first

INTERVENTIONS:
Procedure: Strategy : Supine first — The initial withdrawal in each of 4 segments of the colon: 1)Caecum, Ascending colon and Hepatic flexure 2) Transverse colon 3) Splenic flexure and descending colon 4) Sigmoid colon, will be performed in two different positions. The intervention in this arm will be withdrawal in the supine position and then with dynamic position change.
  Other Names: Dynamic position change; Supine position
  Arms: Strategy : supine first
Procedure: Strategy : dynamic first — The initial withdrawal in each of 4 segments of the colon: 1)Caecum, Ascending colon and Hepatic flexure 2) Transverse colon 3) Splenic flexure and descending colon 4) Sigmoid colon, will be performed in two different positions. The intervention in this arm will be withdrawal with dynamic position change first followed by the supine position.
  Arms: Strategy : dynamic first

SUMMARY:
This study will compare two strategies for colonoscope withdrawal, using polyp detection as the primary outcome measure, to determine the optimal withdrawal strategy.

Null Hypothesis:

On withdrawal of the colonoscope, examining patients with dynamic position change does not yield more polyps than the supine position.

Alternative Hypothesis:

On withdrawal of the colonoscope, examining the patients with dynamic position change improves polyp detection compared to the supine position.

DETAILED DESCRIPTION:
The identification and removal of polyps has been shown to prevent bowel cancer. Although colonoscopy is the best technique to identify polyps, polyps can be missed even in expert hands. Inspection of the bowel occurs predominantly during colonoscope withdrawal. Tailoring a patients position according to the segment of bowel being examined (dynamic position change) is a technique that has been shown to improve visualisation of the bowel wall and polyp detection. However, changing patient position during colonoscope withdrawal has not been widely accepted in clinical practice. This may be because of a lack of awareness of the literature, a perception that the benefit is negligible and the inconvenience of changing a patients position in addition to the small number of publications demonstrating this to be beneficial. We plan to compare the detection of polyps when colonoscope withdrawal is done with dynamic position change (a planned series of position changes to optimise mucosal visualisation) and the supine position (laid on back). These strategies will be compared by performing a double colonoscope withdrawal; The first withdrawal will be performed either supine or in the dynamic position. This will be followed by a second insertion and withdrawal in the alternative position. The order in which these strategies are performed will be randomised i.e. supine then dynamic or dynamic then supine.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnostic colonoscopy
* Age >40 and <80

Exclusion Criteria:

* Inflammatory bowel disease
* Known polyposis syndrome
* Poor mobility which would limit a patients ability to turn

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Colonic polyps | Patients will be included for the duration of their colonoscopy. This would typically be 30-45 minutes.
  The primary outcome for this study is the presence or absence of polyps, detected during colonoscope withdrawal in either the supine position or with dynamic position change.

SECONDARY OUTCOMES:
Colonic polyps | Patients will be included for the duration of their colonoscopy. This would typically be 30-45 minutes.
  The absolute numbers of polyps, the size of polyps and histological type of polyp detected.
Luminal distension | Patients will be included for the duration of their colonoscopy. This would typically be 30-45 minutes.
  Compare the luminal distension of bowel segments in the supine position and with dynamic position change

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Riley, MB ChB, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] Ball AJ, Johal SS, Riley SA. Position change during colonoscope withdrawal increases polyp and adenoma detection in the right but not in the left side of the colon: results of a randomized controlled trial. Gastrointest Endosc. 2015 Sep;82(3):488-94. doi: 10.1016/j.gie.2015.01.035. Epub 2015 Apr 22. PMID 25910661